CLINICAL TRIAL: NCT04619667
Title: Physiological Effects on Respiratory Drive and Transpulmonary Pressure of a New Interface Combining High-flow Nasal Cannula and Cpap in Patients With Mild-to-moderate Acute Respiratory Distress Syndrome: a Pilot Study
Brief Title: Effects of a New Interface for NIV on Respiratory Drive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Prof, University Magna Graecia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OptiPAP Pes
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Acute Respiratory Failure
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High flow nasal cannula (HFNC) (Active Comparator): HFNC will be applied by means of a dedicated device (AIRVO2, Fisher & Paykel Healthcare, Auckland, New Zealand). Gas flow will be set at 50 L/min, and humidification chamber will be set at 31°C.
  Interventions: Device: High Flow Nasal Cannula (HFNC)
- Continuous Positive Airway Pressure (CPAP) (Active Comparator): CPAP will be delivered through a helmet (Castar Next, Intersurgical S.p.A., Mirandola, Italy), with an adjustable Positive End-Expiratory Pressure (PEEP) valve (2.5-20 cmH2O) set at 10 cmH2O (Intersurgical S.p.A., Mirandola, Italy). The helmet will be connected to a turbine-driven ventilator (Monnal T60, Air Liquide Medical Systems, Antony, France) set to deliver oxygen-air admixture at a continuous flow rate of 60 L/min, in order to improve CO2 wash out. No heated humidification will be applied to avoid the "fog effect" in the helmet.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- HFNC+CPAP (Active Comparator): HFNC+CPAP consists in the contemporaneous application of HFNC and CPAP through helmet. HFNC will be set at 30 L/min, with a temperature at 31° C and 100% of relative humidity, while CPAP will be delivered through a helmet (Castar Next, Intersurgical S.p.A., Mirandola, Italy), with an adjustable Positive End-Expiratory Pressure (PEEP) valve (2.5-20 cmH2O) set at 10 cmH2O (Intersurgical S.p.A., Mirandola, Italy). The helmet will be connected to a turbine-driven ventilator (Monnal T60, Air Liquide Medical Systems, Antony, France) set to deliver oxygen-air admixture at a continuous flow rate of 60 L/min, in order to improve CO2 wash out. No heated humidification will be applied to avoid the "fog effect" in the helmet
  Interventions: Device: High Flow Nasal Cannula (HFNC); Device: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Device: High Flow Nasal Cannula (HFNC) — HFNC will be set at 30 L/min, with a temperature at 31° C and 100% of relative humidity
  Arms: HFNC+CPAP; High flow nasal cannula (HFNC)
Device: Continuous Positive Airway Pressure (CPAP) — CPAP will be delivered through a helmet (Castar Next, Intersurgical S.p.A., Mirandola, Italy), with an adjustable Positive End-Expiratory Pressure (PEEP) valve (2.5-20 cmH2O) set at 10 cmH2O (Intersurgical S.p.A., Mirandola, Italy). The helmet will be connected to a turbine-driven ventilator (Monnal T60, Air Liquide Medical Systems, Antony, France) set to deliver oxygen-air admixture at a continuous flow rate of 60 L/min, in order to improve CO2 wash out. No heated humidification will be applied to avoid the "fog effect" in the helmet
  Arms: Continuous Positive Airway Pressure (CPAP); HFNC+CPAP

SUMMARY:
This pilot physiologic randomized cross-over study was designed to investigate if, in patients with hARF, a new device combining high-flow oxygen through nasal cannula (HFNC) and continuous positive airway pressure (CPAP) reduces the respiratory effort, as compared to HFNC and CPAP alone (first outcome). Furthermore, the diaphragm activation, as assessed with ultrasound, gas exchange and patient's comfort among different settings will be assessed (secondary outcomes).

DETAILED DESCRIPTION:
Around 30% of patients admitted to the Intensive Care Unit (ICU) are affected by hypoxemic Acute Respiratory Failure (hARF). The primary supportive treatment in hypoxemic patients is oxygen therapy, which is commonly delivered through nasal prongs or masks. New devices, able to deliver high-flow gas through a nasal cannula (HFNC), have been recently made available. HFNC delivers heated and humidified gas up to 60 L/min, with a fraction of inspired oxygen (FiO2) ranging from 0.21 to 1, via a wide bore soft nasal prong. Warming and humidification of the inspired gas prevent the adverse effects of cool dry gases on the airway epithelium and facilitate expectoration. HFNC also washes out exhaled carbon dioxide (CO2) from the pharyngeal dead space. HFNC has been shown an effective means to deliver oxygen therapy in many clinical conditions.

In healthy subject during spontaneous unassisted breathing, end-expiratory pharyngeal pressure is about 0.3 and 0.8 cmH2O, with open and closed mouth, respectively. Compared to unassisted spontaneous breathing, HFNC generates greater pharyngeal pressure during expiration, while in the course of inspiration it drops to zero, which limits the effectiveness of HFNC in patients with lung edema and/or collapse. By recruiting lung atelectatic regions, reducing venous admixture and decreasing the inspiratory effort, continuous positive airway pressure (CPAP) is likely more effective in these instances. Compared to noninvasive ventilation by application of an inspiratory pressure support, CPAP offers several advantages, which include ease of use and lack of patient-ventilator asynchrony.

CPAP may be applied either through mask or helmet. This latter is better tolerated than facial masks and allows more prolonged continuous CPAP application. When applying CPAP by helmet, however, heating and humidification of the inhaled gas is problematic because of condensation of water inside the interface, so called "fog effect". Moreover, in patients receiving CPAP by helmet some re-breathing occurs.

To overcome these limitations and combine the beneficial effects of HFNC and CPAP, the investigators designed a new device combining HFNC and helmet CPAP.

Recently, this combination was shown to be capable to provide a stable CPAP and effective CO2 washout from the upper airways with negligible CO2 re-breathing. Nonetheless, because of the complex interplay between CPAP and HFNC, the amount of truly applied airway pressure, diaphragm function and temperature inside the helmet might be affected to some extent. In 14 adult healthy volunteers, we found that adding HFNC to CPAP (as referenced to CPAP), 1) did not importantly alter either the pre-set airway pressure during inspiration or temperature inside the helmet; 2) increased expiratory airway pressure proportionally to the flow administered by HFNC, but to a lower extent than HFNC alone (as referenced to spontaneous breathing); 3) determined only slight modifications of the respiratory drive (as assessed through diaphragm ultrasound), compared to CPAP alone, 4) did not cause "fog effect" inside the helmet and 5) did not worsen comfort. We therefore suggested that adding heated humidified air through nasal cannula at a flow of 30 L/min during CPAP would probably be the best setting to be applied in patients with hypoxemic acute respiratory failure.

In patients with hARF, the use of noninvasive respiratory support (CPAP and non-invasive ventilation) is still debated. Patients receiving oxygen therapy, HFNC or CPAP/NIV maintain spontaneous breathing, which allows avoidance of sedation, thus limiting diaphragm dysfunction and delirium, permits easier mobilisation and prevents infections and ICU-acquired weakness. However, the maintenance of spontaneous breathing in patients with damaged lungs and high respiratory drive may result in global/regional pressure/volume changes possibly aggravating initial lung injury. This condition has been defined as patient self-inflicted lung injury (P-SILI). Indeed, respiratory drive is increased in patients with hARF. The high respiratory effort is one of the major determinants of increased transpulmonary pressure (Pl), which is the pressure acting across the lung. Pl represents the pressure alveoli are exposed to, and is considered among the most important determinants of P-SILI. Therefore, the reduction of Pl, across a decrease of the respiratory effort, might be advantageous in patients with hARF.

Investigators have therefore designed this pilot physiologic randomized cross-over study to investigate if, in patients with hARF, HFNC+CPAP reduces the respiratory effort, as compared to HFNC and CPAP (first outcome). Furthermore, we will assess the diaphragm activation, as assessed with ultrasound, gas exchange and patient's comfort among different settings (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* presence of hypoxemic Acute Respiratory Failure, as defined by a respiratory rate greater than 25 breaths/min, an acute onset (within 1 week) of respiratory distress, an arterial oxygen tension (PaO2) and inspiratory oxygen fraction (FiO2) ratio (PaO2/FiO2) lower than 200 mmHg during HFNC, an evidence of bilateral pulmonary infiltrates in the chest X-ray or computed tomography scan, and an absence of history of chronic respiratory failure or moderate-to-severe cardiac insufficiency (New York Heart Association greater than grade 2 or left ventricular ejection fraction <50%).

Exclusion Criteria:

* reduced level of consciousness, as indicated by a Glasgow Coma Scale < 12
* severe respiratory distress (i.e. respiratory rate > 35 breaths/min)
* hemodynamic instability, (i.e. systolic arterial pressure <90 mmHg or mean systolic pressure <65 mmHg despite fluid repletion)
* need for vasoactive agents, i.e. vasopressin or epinephrine at any dosage, or norepinephrine >0.3 mcg/kg/min or dobutamine>5 mcg/kg/min
* life-threatening arrhythmias or electrocardiographic signs of ischemia
* acute respiratory failure secondary to neurological disorders, status asthmaticus, chronic obstructive pulmonary disease (COPD), cardiogenic pulmonary oedema
* presence of tracheotomy
* uncontrolled vomiting
* more than 2 acute organ failures
* body mass index >30 kg/m2
* documented history or suspicion of obstructive sleep apnoea
* contraindications to placement of a nasal-gastric feeding tube
* facial anatomy contraindicating helmet or nasal cannula application
* inclusion in other research protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory effort | After 30 minutes of treatment application
  Inspiratory effort will be assessed as the negative inspiratory swing of the esophageal pressure

SECONDARY OUTCOMES:
Dynamic end-expiratory transpulmonary pressure | After 30 minutes of treatment application
  Difference between airway pressure and end-expiratory esophageal pressure
Dynamic end-inspiratory transpulmonary pressure | After 30 minutes of treatment application
  Difference between airway pressure and end-inspiratory esophageal pressure
Dynamic transpulmonary driving pressure | After 30 minutes of treatment application
  Maximal positive swing in transpulmonary pressure during inspiration
Diaphragm displacement | After 30 minutes of treatment application
  Diaphragm displacement will be assessed with ultrasound to display the cranio-caudal motion of the diaphragm
Diaphragm thickening fraction | After 30 minutes of treatment application
  Thickening fraction will be determined with ultrasound in M-mode at end-expiration (Thickexp) and peak inspiration (Thickinsp) as the distance between the diaphragmatic pleura and the peritoneum
Arterial partial pressure of oxygen (PaO2) | After 30 minutes of treatment application
  Analysis of arterial blood gases
Arterial partial pressure of carbon dioxide (PaCO2) | After 30 minutes of treatment application
  Analysis of arterial blood gases
Patient's comfort | After 30 minutes of treatment application
  It will be measured using an 11-point Numeric Rating Scale. Briefly, after detailed explanation before initiating the protocol, patients will be asked to indicate a number between 0 (worst possible comfort) and 10 (no discomfort) on an adapted printed scale.
Patient's Dyspnea | After 30 minutes of treatment application
  It will be measured using an 11-point Numeric Rating Scale. Briefly, after detailed explanation before initiating the protocol, patients will be asked to indicate a number between 0 (no dyspnoea) and 10 (worst possible dyspnoea) on an adapted printed scale.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Principal Investigator — Magna Graecia University, Anesthesia and Intensive Care Unit

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data will be anonymously shared after reasonable request to the Principal Investigator or Corresponding author
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study and results publication on an international medical journal
Access Criteria: On reasonable request to the corresponding author or principal investigator

REFERENCES:
- [Result] Garofalo E, Bruni A, Pelaia C, Cammarota G, Murabito P, Biamonte E, Abdalla K, Longhini F, Navalesi P. Evaluation of a New Interface Combining High-Flow Nasal Cannula and CPAP. Respir Care. 2019 Oct;64(10):1231-1239. doi: 10.4187/respcare.06871. Epub 2019 Jun 4. PMID 31164484
- [Result] Mauri T, Spinelli E, Mariani M, Guzzardella A, Del Prete C, Carlesso E, Tortolani D, Tagliabue P, Pesenti A, Grasselli G. Nasal High Flow Delivered within the Helmet: A New Noninvasive Respiratory Support. Am J Respir Crit Care Med. 2019 Jan 1;199(1):115-117. doi: 10.1164/rccm.201806-1124LE. No abstract available. PMID 30240275
- [Result] Grieco DL, Menga LS, Raggi V, Bongiovanni F, Anzellotti GM, Tanzarella ES, Bocci MG, Mercurio G, Dell'Anna AM, Eleuteri D, Bello G, Maviglia R, Conti G, Maggiore SM, Antonelli M. Physiological Comparison of High-Flow Nasal Cannula and Helmet Noninvasive Ventilation in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2020 Feb 1;201(3):303-312. doi: 10.1164/rccm.201904-0841OC. PMID 31687831